CLINICAL TRIAL: NCT02914535
Title: A Long-Term Extension Study to Evaluate the Safety of Filgotinib in Subjects With Ulcerative Colitis
Brief Title: Filgotinib in Long-Term Extension Study of Adults With Ulcerative Colitis
Acronym: SELECTIONLTE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-418-3899; 2016-002765-58 (EudraCT Number)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only 3 arms are blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Filgotinib 200 mg (blinded dosing) (Experimental): Filgotinib 200 mg + placebo to match filgotinib 100 mg for up to 336 weeks
  Interventions: Drug: Filgotinib; Drug: Placebo
- Filgotinib 100 mg (blinded dosing) (Experimental): Filgotinib 100 mg + placebo to match filgotinib 200 mg for up to 336 weeks
  Interventions: Drug: Filgotinib; Drug: Placebo
- Placebo (blinded dosing) (Placebo Comparator): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg for up to 336 weeks
  Interventions: Drug: Placebo
- Filgotinib 200 mg (open-label) (Experimental): Filgotinib 200 mg for up to 336 weeks
  Interventions: Drug: Filgotinib
- Filgotinib 100 mg (open-label) (Experimental): Filgotinib 100 mg for up to 336 weeks
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034; GLPG0634
  Arms: Filgotinib 100 mg (blinded dosing); Filgotinib 100 mg (open-label); Filgotinib 200 mg (blinded dosing); Filgotinib 200 mg (open-label)
Drug: Placebo — Tablet(s) administered orally once daily
  Arms: Filgotinib 100 mg (blinded dosing); Filgotinib 200 mg (blinded dosing); Placebo (blinded dosing)

SUMMARY:
The primary objective of this study is to observe the long-term safety of filgotinib in adults who have completed or met protocol specified efficacy discontinuation criteria in a prior filgotinib treatment study in ulcerative colitis (UC).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures associated with this trial
* Must have enrolled in Gilead-sponsored UC parent protocol GS US 418-3898 or any other Gilead/Galapagos-sponsored filgotinib treatment study for UC
* Must have completed all required procedures or met protocol-specified efficacy discontinuation criteria in a prior filgotinib treatment study for UC
* Females of childbearing potential must have a negative pregnancy test at Day 1
* Female individuals of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception for the duration described
* Willingness to refrain from live or attenuated vaccines during the study and for 12 weeks after last dose of study drug

Key Exclusion Criteria:

* Known hypersensitivity to the study drug
* Any chronic medical condition (including, but not limited to, cardiac or pulmonary disease, alcohol or drug abuse) that, in the opinion of the Investigator or sponsor, would make the subject unsuitable for the study or would prevent compliance with the study protocol
* Females of reproductive potential who are unwilling to abide by protocol-specified contraceptive methods as defined
* Use of prohibited medications as outlined in the protocol

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1173 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Overall Safety Profile of Filgotinib Evaluated by Proportion of Participants Experiencing Adverse Events and Abnormal Clinical Laboratory Tests | Up to 336 weeks plus 30 days

SECONDARY OUTCOMES:
Change From Baseline in Components of Mayo Clinic Score (MCS) | Baseline and up to 336 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (323):
- United States (57):
  - Digestive Health Specialists Of The Southeast, Dothan, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - VA Long Beach Healthcare System, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - South Denver Gastroenterology, PC, Lone Tree, Colorado
  - Connecticut GI PC-Research Division, Farmington, Connecticut
  - UF Clinical Research Center, Gainesville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Tampa General Hospital, Tampa, Florida
  - Florida Medical Clinic, P.A, Zephyrhills, Florida
  - Gastroenterology Associates Of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Atlanta Gastroenterology Specialist, PC, Suwanee, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Clinical Trials Unit, Louisville, Kentucky
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital - Crohn's and Colitis Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health Research, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NY Scientific, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Carolina's GI Research LLC, Raleigh, North Carolina
  - Fargo Gastroenterology and Hepatology Clinic, Fargo, North Dakota
  - Consultants for Clinical Research, Cincinnati, Ohio
  - UC Health Physicians Clifton, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine - Baylor Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - TDDC San Marcos, San Marcos, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Spring Gastroenterology, The Woodlands, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Argentina (2):
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata
  - Instituto Médico Cer, Quilmes
- Australia (10):
  - Monash Medical Centre, Clayton, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Coastal Digestive Health, Mountain Creek, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Footscray Hospital, Footscray, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Universitatsklinik Innsbruck, Innsbruck
  - AKH-Medizinische Universitat Wien, Vienna
- Belgium (4):
  - GZA Ziekenhuizen, campus Sint-Vincentius, Antwerp
  - CUB Hopital Erasme, Brussels
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Chretien (CHC) - Clinique Saint-Joseph, Liège
- Bulgaria (3):
  - MHAT Sveti Pantaleymon- Pleven OOD, Pleven
  - "MDHAT Dr. St.Cherkezov" AD, Veliko Tarnovo
  - MHAT "Sveta Petka" AD, Vidin
- Canada (5):
  - University of Calgary, Heritage Medical Research Clinic, Calgary, Alberta
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Hamilton Health Sciences Corporation, McMaster University Medical Centre, Hamilton, Ontario
  - Toronto Digestive Disease Associates Inc., Vaughan, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- Croatia (2):
  - Clinical Hospital Dubrava, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (4):
  - Hepato-Gastroenterology HK, s.r.o., Hradec Králové
  - Oblastni nemocnice Mlada Boleslav, a.s., nemocnice Stredoceskeho kraje, Gastroenterologicke oddeleni, Mladá Boleslav
  - G.E.P. Clinic, s r.o., Prague
  - ISCARE a.s. (Klinicke centrum ISCARE), Klinicke a vyzkumne centrum pro strevni zanety, Prague
- France (18):
  - CHU Amiens Picardie, Amiens
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand - Hopital d'Estaing, Clermont-Ferrand
  - APHP - Hopital Beaujon - Clichy - Universite Paris VII, Clichy
  - CHU de Dijon Bourgogne - Hopital Francois Mitterand, Dijon
  - CHU Grenoble Alpes, La Tronche
  - Hopital Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hopital Nord, Marseille
  - CHU de Montpellier-Hopital Saint Eloi, Montpellier
  - CHU Hotel-Dieu, Nantes
  - Hopital de l'Archet 2, Nice
  - CHU de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - CHU de Saint Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - CHU de Nancy - Hopital Brabois Adultes, Vandœuvre-lès-Nancy
- Georgia (2):
  - Unimed Ajara LLC - Batumi Referral Hospital, Batumi
  - Medi Club Georgia LLC, Tbilisi
- Germany (18):
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - DRK Kliniken Berlin - Westend - Klinik fuer Innere Medizin, Berlin
  - Stadtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitaetsklinik Koln, Cologne
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Westklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Universitatsklinikum Jena, Jena
  - EUGASTRO GmbH, Leipzig
  - Klinikum Luneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitat Munchen - Grosshadern, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitatsklinikum Ulm, Zentrum Fur Innere Medizin, Ulm
- General Hospital of Athens "Hippokratio", 2nd Internal Medicine Clinic of Athens University, Hepato-gastroenterology Unit, Athens, Greece
- Hong Kong (3):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Department of Medicine & Therapeutics, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin
- Hungary (6):
  - Bekes Megyei Kosponti Korhaz, Dr. Rethy Pal Tagkorhaz, IV. Belgyogyaszat - 2. Gasztroenterologia, Békéscsaba
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Kozponti Felnott Szakrendelo, Budapest
  - Szent Janos Korhaz es Eszak-budai Egitett Korhazak, I. Belgyogyaszati - Gasztroenterologiai Osztaly, Budapest
  - Debreceni Egyetem Klinikai Kozpont, II. sz. Belgyogyaszati Klinika, Gasztroenterologia, Debrecen
  - Bugat Pal Korhaz, Belgyogyaszat, Gyöngyös
  - Karolina Korhaz es Rendelointezet, Altalanos Belgyogyaszat-Gasztroenterologia, Mosonmagyaróvár
- India (21):
  - Kaizen Hospital, Ahmedabad
  - M S Ramaiah Medical College and Hospital, Bangalore
  - Apollo Speciality Hospital, Chennai
  - VGM Hospital Institute of Gastroenterology, Coimbatore
  - Gleneagles Global Hospitals, Hyderabad
  - Citizens Specialty Hospital, Hyderabad
  - Centre for Liver Research & Diagnostics, Hyderabad
  - SR Kalla Memorial Gastro and General Hospital, Jaipur
  - S.M.S Medical College & Hospitals, Jaipur
  - Dayanand Medical College & Hospital, Ludhiana
  - Kasturba Medical College (KMC) Hospital, Mangaluru
  - Lokmanya Tilak Municipal General Hospital, Mumbai
  - Midas Multispeciality Hospital Pvt. Ltd, Nagpur
  - Suretech Hospital & Research Centre Ltd, Nagpur
  - Grant Medical Foundation Ruby Hall Clinic, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Gandhi Hospital, Secunderabad
  - Surat Institute of Digestive Sciences, Surat
  - Kasturba Hospital Medical College, Udupi
  - Sterling Hospital, Vadodara
  - Samvedna Hospital, Varanasi
- Beaumont Hospital, Dublin, Ireland
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (8):
  - UOC Gastroenterologia II, Castellana Grotte
  - U.O. Fisiopatologia Digestiva, Catanzaro
  - Ospedale Clinicizzato SS. Annunziata - Dipartimento di Medicina, Chieti
  - Endocsopia Digestiva Centralizzata - ASST Fatebenefratelli Sacco, Ospedale Fatebenefratelli e Oftalmico, Milan
  - UOC Gastroenterologia, Padua
  - Azienda Ospedaliero-Universitaria Pisana - Presidio Ospedaliero Cisanello, Pisa
  - UOC Gastroenterologia ed Endoscopia Digestiva, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (42):
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka University Hospital, Suita, Osaka
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyō City
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital, Chūōku
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Tokai University Hachioji Hospital, Hachiōji
  - Hiroshima University Hospital, Hiroshima
  - Fukuoka University Hospital, Jonan-ku
  - Ofuna Chuo Hospital, Kamakura
  - Kitakyushu City Hospital Organization Kitakyushu Municipal Medical Center, Kitakyushu-shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurume University Hospital, Kurume-shi
  - Hidaka Coloproctology Clinic, Kurume-shi
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - The Jikei University Hospital, Minatoku
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka-shi
  - Iwate Medical University Hospital, Morioka
  - Aichi Medical University Hospital, Nagakute-shi
  - Saiseikai Niigata Daini Hospital, Nishiku
  - Hyogo College of Medicine College Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - Osaka City University Hospital, Osaka
  - Wakakusa-Daiichi Hospital, Osaka
  - Ishida IBD Clinic, Ōita
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga-Ken Medical Centre Koseikan, Saga
  - Saga University Hospital, Saga
  - Kitasato University Hospital,THE KITASATO INSTITUTE, Sagamihara
  - Tokito Clinic, Saitama
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - National Hospital Organization Sendai Medical Center, Sendai
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Osaka Medical College Hospital, Takatsuki
  - Ieda Hospital, Toyota-shi
  - Wakayama Medical University Hospital, Wakayama
  - Colo-proctology Center Matsushima Clinic, Yokohama
- Malaysia (2):
  - Hospital Pulau Pinang, George Town
  - Hospital Queen Elizabeth, Kota Kinabalu
- PCR-Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli, Mexico
- Netherlands (3):
  - Academic Medical Center (AMC), Amsterdam
  - Gelre Hospital, Apeldoorn
  - University Medical Center Utrecht, Utrecht
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Auckland City Hospital, Grafton
  - Wellington Hospital, Newtown
  - Bay of Plenty District Health Board - Tauranga Hospital, Tauranga
- Poland (21):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Gastroenterologii i Chorob Wewnetrznych, Bialystok
  - VITAMED Galaj i Cichomski spólka jawna, Bydgoszcz
  - Gabinet Lekarski Janusz Rudzinski, Bydgoszcz
  - NZOZ INTER-MED, Centrum Endoskopowe, Częstochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej ALL-MEDICUS, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Santa Familia, Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Centrum Innowacyjnych Terapii Sp. z o.o., Piaseczno
  - Clinical Research Center Spolka z ograniczna odpowiedzialnoscia Medic-R Sp. k., Poznan
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów
  - Endoskopia Sp. z o.o., Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Kopon, Zmudzinski i Wspolnicy Sp. j. Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - H-T.Centrum Medyczne Spolka z Ograniczona Odpowiedzialnoscia Sp.K., Tychy
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administacji w Warszawie, Warsaw
  - Niepubliczny Zaklad Opieki Zrodotnej VIVAMED Jadwige Miecz, Warsaw
  - Bodyclinic, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (2):
  - Hospital da Senhora da Oliveira Guimaraes, E.P.E., Guimarães
  - Centro Hospitalar de Sao Joao, EPE, Porto
- Romania (4):
  - MedLife, Gastroenterologie, Bucharest
  - Spitalul Clinic Colentina - Sectia de Spitulal Clinic Colentina, Gastroenterologie, Bucharest
  - Cabinet Medical Individual Dr Tirnaveanue Amelita, Gastroenterologie, Oradea
  - Cabinet Particular Policlinic Algomed SRL, Timișoara
- Russia (14):
  - State Budgetary Healthcare Institution "Chelyabinski Regional Clinical Hospital", Chelyabinsk
  - State Budgetary Institution of Health Irkustsk Order "Badge of Honor" Regional Clinical Hospital, Irkutsk
  - Federal State Budgetary Institution of Science Federal Research Center of Nutrition, Biotechnology and Food Safety, Moscow
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital # 24 of Healthcare Department of Moscow", Moscow
  - State Budgetary Healthcare Institution of Moscow Region "Moscow Regional Clinical Research Institute n.a. M.F. Vladimirskiy", Moscow
  - State Budgetary Healthcare Institution of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a. N.A., Nizhny Novgorod
  - State Budgetary Institution of Health of Novosibirsk Region "City Clinical Hospital #12", Novosibirsk
  - State Budgetary Healthcare Institution of the Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk
  - Saint Petersburg State Budgetary Healthcare Institution "City Polyclinic #38", Saint Petersburg
  - "Riat" LLC, Saint Petersburg
  - "Scientific Research Centre ECO-safety" LLC, Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
  - Treatment and Prevention Interdistrict Institution "Smolenskie kliniki" LLC, Smolensk
  - Tyumen Regional State Autonomous Healthcare Institution << Consulting and Diagnostic Centre <<Endos>>, Tyumen
- Zvezdara University Medical Center, Belgrade, Serbia
- Singapore General Hospital, Singapore, Singapore
- KM Management, s.r.o., Gastroenterologicke a hepatologicke centrum Nitra, Nitra, Slovakia
- South Africa (2):
  - Dr MJ Prins, Cape Town
  - Peermed Clinical Trial Centre, Johannesburg
- South Korea (9):
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Division of Gastroenterology, Department of Medicine, Samsung Medical Center, Seoul
  - Kyung Hee University Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (5):
  - Centro Medico Teknon, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocío, Seville
- Sweden (3):
  - Skane University Hospital, Malmo
  - Danderyd University Hospital Corp, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - Gastroenterologische Praxis Balsiger, Seibold und Partner, Bern
  - Universitätsspital Zürich, Zurich
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District
- Ukraine (17):
  - Municipal Institution "Cherkasy Regional Hospital of Cherkasy Regional Council", Gastroenterology Department, Cherkasy
  - Municipal City Clinical Hospital of the Emergency Medical Care, 1 st Therapy Department. Danylo Halytsky Lviv National Medical, Chernivtsi
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", Surgical Department, Chernivtsi
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipropetrovsk
  - Ivanto-Frankivsk Central City Clinic Hospital, Therapy Department #1. State Higher Education Institution Ivano-Frankivsk National, Ivano-Frankivsk
  - Municipal Health Care Institution "Kharkiv City Clinical Hospital #2 named after prof. O. O. Shalimov", Proctology Department, Kharkiv
  - L.T. Mala State Institution "National Institute of Therapy of National Academy of Medical Sciences of Ukraine", Kharkiv
  - Municipal Institution of Health Care "Regional Hospital of War Veterans", Therapeutic Department No1, Kharkiv
  - Kyiv City Clinical Hospital No. 18, Proctology Department, Kyiv
  - Municipal Non-profit Enterprise "Consultative and Diagnostic Center" of Pechersk District of Kyiv, Therapy Department, Kyiv
  - Odesa Clinical Railway Hospital Branch of "Healthcare Center" of Public joint stock company "Ukrainian Railway", Odesa
  - Municipal Institution "Odesa Regional Clinical Hospital", Regional Gastroenterology Center based on Surgery Department, Odesa
  - Ternopil University Hospital, Regional Center of Gastroenterology with Hepatology, Ternopil
  - Vinnytsia Regional Clinical Hospital of War Veterans, Therapy Department #1, Vinnytsia
  - M.I. Pyrogov Vinnytsia Regional Clinical Hospital, Gastroenterology Department, Vinnytsia
  - Medical Center LLC "Health Clinic", Vinnytsia
  - Municipal Institution "Zaporizhzhya Regional Clinical Hospital" of Zaporizhzhya Regional Council, Zaporizhzhya
- United Kingdom (13):
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, Norfolk
  - The Pennine Acute Hospitals NHS Trust, Bury
  - Cambridge University Hospital NHS Foundation Trust, Cambridge
  - Royal Derby Hospital, Derby
  - NHS Lothian, Edinburgh
  - Glasgow Clinical Research Facility - Queen Elizabeth University Hospital, Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Wycombe Hospital, High Wycombe
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, London
  - Biomedical Research Unit, Nottingham
  - Oxford University Hospitals NHS Trust, Oxford
  - St Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - Southampton National Institute for Health Research, Wellcome Trust Clinical Research Facility, Southampton

REFERENCES:
- [Derived] Feagan BG, Matsuoka K, Rogler G, Laharie D, Vermeire S, Danese S, Loftus EV Jr, Beales I, Schreiber S, Kim HJ, Faes M, de Haas A, Masior T, Rudolph C, Peyrin-Biroulet L. Long-term safety and efficacy of filgotinib for the treatment of moderately to severely active ulcerative colitis: Interim analysis from up to 4 years of follow-up in the SELECTION open-label long-term extension study. Aliment Pharmacol Ther. 2024 Sep;60(5):563-584. doi: 10.1111/apt.18158. Epub 2024 Jul 31. PMID 39086130
- [Derived] Schreiber S, Rogler G, Watanabe M, Vermeire S, Maaser C, Danese S, Faes M, Van Hoek P, Hsieh J, Moerch U, Zhou Y, de Haas A, Rudolph C, Oortwijn A, Loftus EV Jr. Integrated safety analysis of filgotinib for ulcerative colitis: Results from SELECTION and SELECTIONLTE. Aliment Pharmacol Ther. 2023 Nov;58(9):874-887. doi: 10.1111/apt.17674. Epub 2023 Sep 18. PMID 37718932
- [Derived] Vermeire S, Feagan BG, Peyrin-Biroulet L, Oortwijn A, Faes M, de Haas A, Rogler G. Withdrawal and Re-treatment with Filgotinib in Ulcerative Colitis: Post Hoc Analyses of the Phase 2b/3 SELECTION and SELECTIONLTE Studies. J Crohns Colitis. 2024 Jan 27;18(1):54-64. doi: 10.1093/ecco-jcc/jjad123. PMID 37540206